CLINICAL TRIAL: NCT00003636
Title: A Randomized Phase III Study Comparing Upfront Debulking Surgery Versus Neo-Adjuvant Chemotherapy in Patients With Stage IIIC or IV Epithelial Ovarian Carcinoma
Brief Title: Chemotherapy Plus Surgery in Treating Patients With Stage III or Stage IV Ovarian, Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-55971; EORTC-55971
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Cisplatin; Neoadjuvant Therapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining surgery with chemotherapy may kill more tumor cells. It is not yet known whether chemotherapy before surgery is more effective than chemotherapy after surgery in treating ovarian, peritoneal, or fallopian tube cancer.

PURPOSE: This randomized phase III trial is studying chemotherapy given before surgery to see how well it works compared to chemotherapy given after surgery with or without additional surgery in treating patients with stage III or stage IV ovarian cancer, peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and progression-free survival in patients with stage IIIC or IV ovarian epithelial, peritoneal, or fallopian tube carcinoma treated with neoadjuvant chemotherapy followed by interval debulking surgery versus upfront cytoreductive surgery followed by chemotherapy with or without interval debulking surgery.
* Compare the quality of life of patients treated with these regimens.
* Compare the different treatment complications in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, method of biopsy, stage, largest tumor size before surgery, and intent to also randomize on EORTC-55012. Patients are randomized to one of two treatment arms.

* Arm I: Patients undergo upfront maximal cytoreductive surgery followed by cisplatin or carboplatin IV every 3 weeks for 3 courses. Patients with non-optimal primary debulking may undergo interval debulking surgery at the physician's discretion. All patients then receive an additional 3 courses of the same regimen of chemotherapy.
* Arm II: Patients receive chemotherapy as in arm I. Patients with stable or responding disease undergo interval debulking surgery followed by an additional 3 courses of the same regimen of chemotherapy.

Second-look surgery is allowed for both arms if clinically indicated.

Quality of life (QOL) is assessed prior to treatment, after the third and sixth course of chemotherapy, and at 6 and 12 months after study. Patients who are also randomized on EORTC-55012 follow the QOL assessment schedule for EORTC-55012 only.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 704 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IIIC or IV ovarian epithelial carcinoma, peritoneal carcinoma, or fallopian tube carcinoma

  * If biopsy is not available, evidence of adenocarcinoma by fine needle aspiration allowed if all of the following are true:

    * Presence of pelvic ovarian mass
    * Omental cake or other metastasis larger than 2 cm in the upper abdomen and/or regional lymph node metastasis
    * CA 125/carcinoembryonic antigen ratio greater than 25 (if ratio less than 25, barium enema or colonoscopy AND gastroscopy or radiological examination of the stomach must be negative for primary tumor)
    * Normal mammography (if CA 125/carcinoembryonic antigen ratio less than 25)
* Tumor greater than 2 cm, excluding ovaries, on laparoscopy or CT scan
* No brain or leptomeningeal metastases

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.25 times upper limit of normal (ULN)

Renal:

* Creatinine less than 1.25 times ULN

Other:

* No other serious disabling diseases contraindicating primary cytoreductive surgery or primary platin-based chemotherapy
* No other prior primary malignancies except carcinoma in situ of the cervix or basal cell carcinoma of the skin
* No psychological, familial, sociological, or geographical condition potentially preventing protocol compliance or follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No other prior procedures except diagnostic biopsy by laparotomy or laparoscopy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 1998-09; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Overall survival as measured by Kaplan Meier every 3 months for 2 years, every 6 months for 3 years, and then annually

SECONDARY OUTCOMES:
Progression-free survival as measured by Kaplan Meier and RECIST every 3 months for 2 years, every 6 months for 3 years, and then annually
Health-related quality of life as measured by Quality of Life Questionnaire-C30 after courses 1, 3 and 6, then at 6 and 12 months
Toxicity as measured by NCIC Common Toxicity Criteria v2.0 within 4 weeks of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ignace B. Vergote, MD, PhD, Study Chair — U.Z. Gasthuisberg, Leuven
Locations (65):
- Argentina (2):
  - Hospital de Clinicas "Jose De San Martin", Buenos Aires
  - Shaare Zedek Medical Center, Buenos Aires
- Austria (4):
  - Karl-Franzens-University Graz, Graz
  - Innsbruck Universitaetsklinik, Innsbruck
  - Allgemeines Krankenhaus - Universitatskliniken, Vienna
  - Ludwig Boltzmann Institute for Applied Cancer Research at Kaiser Franz Josef Hospital, Vienna
- Belgium (4):
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - U.Z. Gasthuisberg, Leuven
- Canada (12):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
- Herlev Hospital - University Hospital of Copenhagen, Copenhagen, Denmark
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Institut Claudius Regaud, Toulouse
- Martin Luther Universitaet, Halle, Germany
- Ireland (2):
  - Coombe Women's Hospital, Dublin
  - St. James's Hospital, Dublin
- Italy (5):
  - Spedali Civili di Brescia, Brescia
  - Mirano General Hospital, Mirano-Venice
  - Libero Istituto Universitario Campus Bio-Medico, Rome
  - Azienda Sanitaria Ospedaliera Ordine Mauriziano, Torino
  - Clinica Universitaria, Turin
- Netherlands (8):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Akademisch Ziekenhuis Vrije Universiteit - Medisch Centrum, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - Erasmus MC - Sophia Children's Hospital, Rotterdam
- Norway (2):
  - Haukeland Hospital - University of Bergen, Bergen
  - Norwegian Radium Hospital, Oslo
- Portugal (2):
  - Hospitais da Universidade de Coimbra (HUC), Coimbra
  - Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon
- Spain (4):
  - Institut d'Oncologia Corachan, Barcelona
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
- Sweden (4):
  - Lund University Hospital, Lund
  - Karolinska University Hospital - Huddinge, Stockholm
  - Umea Universitet, Umeå
  - Uppsala University Hospital, Uppsala
- United Kingdom (10):
  - Royal United Hospital, Bath, England
  - Cheltenham General Hospital, Cheltenham, England
  - University College of London Hospitals, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Staffordshire General Hospital, Stafford, England
  - Western Infirmary, Glasgow, Scotland
  - Queen Elizabeth The Queen Mother Hospital, Margate

REFERENCES:
- [Background] Chi DS, Musa F, Dao F, Zivanovic O, Sonoda Y, Leitao MM, Levine DA, Gardner GJ, Abu-Rustum NR, Barakat RR. An analysis of patients with bulky advanced stage ovarian, tubal, and peritoneal carcinoma treated with primary debulking surgery (PDS) during an identical time period as the randomized EORTC-NCIC trial of PDS vs neoadjuvant chemotherapy (NACT). Gynecol Oncol. 2012 Jan;124(1):10-4. doi: 10.1016/j.ygyno.2011.08.014. Epub 2011 Sep 13. PMID 21917306
- [Result] Verleye L, Ottevanger PB, Kristensen GB, Ehlen T, Johnson N, van der Burg ME, Reed NS, Verheijen RH, Gaarenstroom KN, Mosgaard B, Seoane JM, van der Velden J, Lotocki R, van der Graaf W, Penninckx B, Coens C, Stuart G, Vergote I. Quality of pathology reports for advanced ovarian cancer: are we missing essential information? An audit of 479 pathology reports from the EORTC-GCG 55971/NCIC-CTG OV13 neoadjuvant trial. Eur J Cancer. 2011 Jan;47(1):57-64. doi: 10.1016/j.ejca.2010.08.008. Epub 2010 Sep 16. PMID 20850296
- [Result] Vergote I, Trope CG, Amant F, Kristensen GB, Ehlen T, Johnson N, Verheijen RH, van der Burg ME, Lacave AJ, Panici PB, Kenter GG, Casado A, Mendiola C, Coens C, Verleye L, Stuart GC, Pecorelli S, Reed NS; European Organization for Research and Treatment of Cancer-Gynaecological Cancer Group; NCIC Clinical Trials Group. Neoadjuvant chemotherapy or primary surgery in stage IIIC or IV ovarian cancer. N Engl J Med. 2010 Sep 2;363(10):943-53. doi: 10.1056/NEJMoa0908806. PMID 20818904
- [Result] Fruehauf JP, Yu I, Parker R: In vitro drug response and biomarker profiles for ovarian cancer specimens obtained at initial debulking or after neoadjuvant chemotherapy (EORTC 55971). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2177, 2002.
- [Derived] Tajik P, van de Vrie R, Zafarmand MH, Coens C, Buist MR, Vergote I, Bossuyt PMM, Kenter GG. The FIGO Stage IVA Versus IVB of Ovarian Cancer: Prognostic Value and Predictive Value for Neoadjuvant Chemotherapy. Int J Gynecol Cancer. 2018 Mar;28(3):453-458. doi: 10.1097/IGC.0000000000001186. PMID 29324537
- [Derived] Vizzielli G, Fanfani F, Chiantera V, Tortorella L, Lucidi A, Petrillo M, Costantini B, Scambia G, Fagotti A. Does the diagnosis center influence the prognosis of ovarian cancer patients submitted to neoadjuvant chemotherapy? Anticancer Res. 2015 May;35(5):3027-32. PMID 25964591
- [Derived] van Meurs HS, Tajik P, Hof MH, Vergote I, Kenter GG, Mol BW, Buist MR, Bossuyt PM. Which patients benefit most from primary surgery or neoadjuvant chemotherapy in stage IIIC or IV ovarian cancer? An exploratory analysis of the European Organisation for Research and Treatment of Cancer 55971 randomised trial. Eur J Cancer. 2013 Oct;49(15):3191-201. doi: 10.1016/j.ejca.2013.06.013. Epub 2013 Jul 11. PMID 23850170